CLINICAL TRIAL: NCT01821885
Title: Effectiveness of Spirometry and the Report of Spirometric Test Results by a Primary Care Physician on Smoking Cessation Rate in Adult Smokers: a Randomized Controlled Trial.
Brief Title: Effectiveness of Spirometry as a Motivational Tool to Quit Smoking
Acronym: ESPIMOAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Mº Isabel Irizar Aramburu, family doctor, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011111013; KRONIK11/071 - EJGV 2011111013 (Other: KRONIKGUNE - EUSKO JAURLARITZA/GOBIERNO VASCO)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Smoking Cessation; COPD
Keywords: Spirometry; screening; smoking cessation; tobacco; COPD
MeSH Terms: conditions — Smoking Cessation; Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Spirometry and a brief advice to quit smoking (Experimental): Intervention group:
  The intervention consists of completing a questionnaire and undergo spirometry with bronchodilator test by a trained nurse. Later, the patients receives a brief advice to quit smoking and a report of the spirometry results by their family doctor.
  Interventions: Behavioral: Spirometry and a brief advice to quit smoking
- Brief advice to quit smoking (Active Comparator): Control group:
  Patients in the control group complete a questionnaire by a nurse and then receive a brief advice to quit smoking by their family doctor.
  Interventions: Behavioral: Brief advice to quit smoking

INTERVENTIONS:
Behavioral: Spirometry and a brief advice to quit smoking — During a year, recruitment for active smoker patients was done by doctors in primary care medical offices. In the intervention group, after been randomized, one trained nurse completed the questionnaires and did the spirometry with bronchodilator test and set a date with its family doctor who did a minimal smoking cessation counselling intervention and informed the patients about the spirometry results according to established protocol.
  Arms: Spirometry and a brief advice to quit smoking
Behavioral: Brief advice to quit smoking — During a year, recruitment for active smokers patients occurred through doctors in primary care medical offices. After be randomized, in de control group, a nurse complete the questionnaires. Below, patients go to the family doctor who will do a minimal smoking cessation counselling intervention.
  Arms: Brief advice to quit smoking

SUMMARY:
The aim of the study is to asses the efficacy of the spirometry and a minimal smoking cessation counselling intervention to quit smoking after a year in patients older than 40 years, smokers of more than 10 packs-year and without a chronic obstructive pulmonary disease (COPD) diagnosis.

ELIGIBILITY:
Inclusion Criteria:

- Active smokers over 40 years and more than 10 pack-years

Exclusion Criteria:

* Previous diagnosis of respiratory disease (asthma, COPD, interstitial lung disease) that cause alteration of spirometric pattern.
* Patients with limitations in performing spirometry
* Age greater than 80 years
* Institutionalized patients
* Patients with a life expectancy less than 1 year
* Spirometry in the past 2 years

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary measure of results will be the differences in smoking cessation rates between intervention and control groups | 12 months after been conducted the intervention
  In all patients who report smoking withdrawal, smoking cessation will be confirmed by air carbon monoxide concentration.

SECONDARY OUTCOMES:
Reduce the number of cigarettes among those who continue smoking | 12 months after been conducted the intervention
  One secondary outcome will be to reduce the number of cigarettes. In all patients who continue smoking will be recorded the number of cigarettes smoked per day currently
Increase smoking abstinence rates in patients with COPD | 12 months after been conducted the intervention
  Evaluate the differences in smoking cessation rates between patients with COPD and those without.

CONTACTS AND LOCATIONS:
Overall Officials: Mª Isabel Irizar Aramburu, Principal Investigator — Osakidetza
Locations (1):
- Basque health service, Vitoria-Gasteiz, Alava 45, Spain

REFERENCES:
- [Derived] Irizar-Aramburu MI, Martinez-Eizaguirre JM, Pacheco-Bravo P, Diaz-Atienza M, Aguirre-Arratibel I, Pena-Pena MI, Alba-Latorre M, Galparsoro-Goikoetxea M. Effectiveness of spirometry as a motivational tool for smoking cessation: a clinical trial, the ESPIMOAT study. BMC Fam Pract. 2013 Dec 5;14:185. doi: 10.1186/1471-2296-14-185. PMID 24308728